CLINICAL TRIAL: NCT03627962
Title: Using Gaze-directed Oculomotor Training (GDOMT) to Enhance Reading-related Oculomotor Skills and Chinese Characters Recognition CCR) for Children With Neuromuscular Disease (NMD)
Brief Title: Oculomotor Training and Chinese Characters Recognition in Children With Neuromuscular Disease
Acronym: yes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Carly Lam, Principal investigator, Professor Carly SY Lam, PHD, Associate Dean of Faculty of Health and Social Sciences, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSEARS20160816001
Record Dates: First submitted 2018-03-27; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Extraocular Muscle Disorder; Neuromuscular Diseases
Keywords: gaze-directed oculomotor training, reading in Chinese
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gaze-directed oculomotor training (Experimental): device: Tobii PCEye Treatment group went through the oculomotor training with a gaze-pointer interface (Tobii PC Eye) in reading in Chinese.
  Interventions: Other: gaze-directed oculomotor training
- control (No Intervention): No intervention: participants in control read ordinary Chinese textbooks.

INTERVENTIONS:
Other: gaze-directed oculomotor training — Device: Tobii PCEye
  Protocol: Visual span was calculated by the distance between human-computer and dpi of fonts. Pointer speed was programmed 120pixels (5 degrees)/1sec for image drift of reading.
  Dosage: 1) gaze-access required 20 to 10 degrees per fixation to activate text-to-speech (TTS) read-aloud function; about 30 repetitions of saccade and fixation.
  2) gaze-directed OMT limited to 10-5 degrees. Chinese characters recognition in multiple choice format, about 60 repetitions.
  Target behavior - gaze-directed access by Tobii PCEye: reading from left to right (=horizontal mouse mover); read-aloud function by gaze dwell > 500ms. To enhance purposeful and repetitive eye movement.
  Frequency: 2 session/wk x 8 wks
  Duration: 30 min/session
  Other Names: Tobii PCEye
  Arms: gaze-directed oculomotor training

SUMMARY:
The aim of this study is to investigate the effects of gaze-directed oculomotor training incorporated with web-based curriculum readings in Chinese to enhancing fixation, saccade and Chinese characters recognition in schoolchildren with neuromuscular disease associated with congenital oculomotor anomalies.

DETAILED DESCRIPTION:
Background: schoolchildren with neuromuscular diseases associated with congenital oculomotor anomalies find problems in reading, even found difficulties in learning their mother-tongue language of Chinese.

Objectives: (1) To test the hypothesis of using gaze-directed oculomotor training (GDOMT) incorporated with curriculum-based reading platform might enhance reading-related oculomotor skills and Chinese characters recognition; (2) To validate the outcome parameters of reading-related oculomotor skills by using remote eye tracker.

Hypothesis: It has been shown that motor learning theory were effective in motor training for children with neuromuscular diseases. Oculomotor training to re-gain reading skills has been found effective for person with acquired brain injury or children with dyslexia, but there is no study on oculomotor training in children with neuromuscular diseases for reading. In this study, we hypothesize that self-initiated gaze-directed oculomotor training via e-reading platform (activated by horizontal saccade from left to right, then fixation dwell about 500ms to activate read-aloud the words phrases in Cantonese) for children with neuromuscular diseases associated with extra-ocular muscles anomalies, will be improved accuracy in fixation and saccade.

Design: Cross-centers prospective Cohort study with quasi-experimental design; subjects of aged 6 to 8, randomly assigned into age-matched treatment group (N=10) or the age-matched control group (N=11).

Methods: Participants (aged 6 to 8) with neuromuscular diseases, ocular health normal, normal intelligence, studying in main-stream special schools for children with physically disabilities were recruited. Participants passed the vision screening then randomized to age-paired matched control group (N=11) and treatment group (N=10). After time 1 measure, they attended reading class as usual. Therapists or teaching staff brought participants to library one by one and let the participant to read hardcopy or e-reading as assigned control or treatment group. Those therapists and teaching staff involved in training did not involve in repeated measures.

Both groups explored to their curriculum-based reading materials. Participants of treatment group received oculomotor training by means of using a gaze-pointer interface to activate a reading e-platform, while control group used some ordinary hardcopy printout as placebo.

Training sessions were provided twice per week for eight consecutive school calendar weeks. Occupational therapists and teachers collaborated in the reading class throughout 8 weeks. Participant in treatment group sat in front of the computer with the access hardware PCEye, gaze-directed oculomotor training was facilitated by decreasing the visual span from 20 to 10 to 5 degrees per words phrase.

Teacher presented the web-based reading materials in hardcopies (placebo) to control group. Teacher pointed to the passages and read aloud to individual. Both treatment group and control group have same dosage of reading.

Control group performed the Chinese characters recognition test by gesture or verbal responses to the printout of web-based materials, while treatment group used gaze-access to select the answers same as Developmental Eye Movement Sub-test C.

ELIGIBILITY:
Inclusion Criteria:

* schoolchildren with neuromuscular disease associated with oculomotor anomalies,
* study in primary school of normal intelligence;
* age 6 to 8 years old;
* with native language in Chinese and Cantonese;
* because of pure oculomotor training, subjects with aphasia may also be recruited;
* students with normal to mild visual impairment (best corrected visual acuity is better than 20/60);and
* both eyes without visual loss as Tobii X3-120 seek binocular vision for calibration and assessment.

Exclusion Criteria:

* students with mild to moderate intellectual disability;
* students unable to read Chinese or unable to understand spoken Cantonese;
* student without oculomotor anomalies who are expected to have accurate fixation and saccades; or student with moderate to severe visual impairment; and
* students with ADHD, ASD or with behaviour challenging and attention problems, and/or with epileptic seizure elicited by computer flickering light.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
adjusted horizontal reading time | 24 weeks
  number of corrected fixation per total visit duration of 80 Area of interest (AOI). It was tested by the Developmental Eye Movement test, subtest C.

SECONDARY OUTCOMES:
saccade accuracy | 24 weeks
  number of correct saccade sequence (5 AOI) per 16 lines
Chinese characters recognition accuracy of grade-leveled readings | 24 weeks
  percentage of correct answer per 10 multiple choice questions, select 1 out of 10

CONTACTS AND LOCATIONS:
Overall Officials: Carly SY Lam, PhD, Study Director — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong